CLINICAL TRIAL: NCT02623192
Title: Respiratory Mechanics in Acute Respiratory Distress Syndrome: A Quality Improvement-based Registry
Brief Title: Respiratory Mechanics Registry for ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Beijing Tiantan Hospital (Other); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: REB# 15-098
Record Dates: First submitted 2015-07-30; First posted 2015-12-07 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ARDS
  Interventions: Other: Patients who have performed the ARDS pulmonary function test

INTERVENTIONS:
Other: Patients who have performed the ARDS pulmonary function test

SUMMARY:
This registry was proposed to investigate the epidemiology of respiratory mechanics in patients with ARDS through collecting data from a QI project which was constituted with systematic assessments of respiratory mechanics and gas exchange.

DETAILED DESCRIPTION:
The amount of respiratory impairment in patients with Acute Respiratory Distress Syndrome (ARDS) is variable and applying the same ventilator regimen to every patient is questionable. In order to individualize ventilator management, monitoring respiratory mechanics may help to decide ventilator settings or set limits. A systematic assessment of respiratory mechanics and gas exchange response in patients who meet the criteria for ARDS has been initiated as a Quality Improvement (QI) project in the Department of Critical Care at St. Michael's Hospital. The QI project aims to facilitate the use of these parameters for ventilatory management. Measurements include: respiratory system, lung and chest wall mechanics (elastance and resistance), oxygenation response to positive end-expiratory pressure (PEEP), and estimate of alveolar recruitability using a simplified bedside maneuver[1]. Placement of an esophageal catheter is considered when the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) ≤200 mmHg[2]. Audits are performed to see whether the measurements influence ventilatory management. Collecting these data into a registry will elicit helpful epidemiological information since the current epidemiological knowledge surrounding respiratory mechanics abnormalities in ARDS is limited. A registry with a large sample size may inform future recommendations. The investigators therefore propose to introduce the collected data from our QI program into an ARDS registry. Similar data obtained from other centers may also contribute to the registry in the future. The primary objective of the registry will be to investigate the epidemiology of abnormal respiratory mechanics in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Medical-Surgical ICU, Trauma-Neuro ICU, and Cardiovascular ICU who meet the Berlin definition of ARDS and receive invasive ventilation.

Exclusion Criteria:

* Severe hemodynamic instability: > 30% variation of mean arterial pressure and/or heart rate (HR) in the last 2 hours or the need for a high dose of vasopressors (higher than 0.5 µg/kg/min of norepinephrine);
* Patients who present with a known esophageal problem, active upper gastrointestinal bleeding, or any other contraindication for the insertion of a gastric tube.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have performed the ARDS pulmonary function test will be eligible for the registry. The clinical team discuss on a case-by-case basis to determine whether an ARDS patient is appropriate to received the ARDS pulmonary function test (systematic assessment of respiratory mechanics in the QI portion)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Driving pressure (centimetre of water) | One hour
  Epidemiology of physiological abnormalities in respiratory mechanics were be reported.

SECONDARY OUTCOMES:
Transpulmonary pressure (centimetre of water) | One hour
Respiratory compliance (millilitre / centimetre of water) | One hour
Lung compliance (millilitre / centimetre of water) | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- St. Michael's Hospital, Toronto, Ontario, Canada
- Catholic University of the Sacred Heart, Rome, Lazio, Italy

REFERENCES:
- [Background] Dellamonica J, Lerolle N, Sargentini C, Beduneau G, Di Marco F, Mercat A, Richard JC, Diehl JL, Mancebo J, Rouby JJ, Lu Q, Bernardin G, Brochard L. PEEP-induced changes in lung volume in acute respiratory distress syndrome. Two methods to estimate alveolar recruitment. Intensive Care Med. 2011 Oct;37(10):1595-604. doi: 10.1007/s00134-011-2333-y. Epub 2011 Aug 25. PMID 21866369
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Derived] Chen L, Chen GQ, Shore K, Shklar O, Martins C, Devenyi B, Lindsay P, McPhail H, Lanys A, Soliman I, Tuma M, Kim M, Porretta K, Greco P, Every H, Hayes C, Baker A, Friedrich JO, Brochard L. Implementing a bedside assessment of respiratory mechanics in patients with acute respiratory distress syndrome. Crit Care. 2017 Apr 4;21(1):84. doi: 10.1186/s13054-017-1671-8. PMID 28372575